CLINICAL TRIAL: NCT06249139
Title: Caring4Caregivers: A Theory-driven Mobile Solution to Promote Self-care and Well-being Among Caregivers of Individuals With Alzheimer's and Related Dementias
Brief Title: Compass for Care: A Theory-driven Mobile Solution to Promote Well-being Among Caregivers of Individuals With ADRD
Acronym: Compass4Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pro-Change Behavior Systems (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R44AG076345 (NIH)
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Dementia; Mental Health
Keywords: Transtheoretical Model; Stages of change; Alzheimer's Disease; Caregiving; Dementia; Well-being
MeSH Terms: conditions — Dementia; Psychological Well-Being; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compass for Care (Well-being intervention) (Experimental): Participants receive 12 weekly modules containing interactive activities and static content and tailored messages delivered via text message or email. The intervention focuses on five self-care behaviors critical to ADRD caregiver well-being: 1) taking time to recharge; 2) finding information about your loved one's diagnosis and needs; 3) discovering your strengths and limits; 4) exploring outside help; and 5) seeking emotional support.
  Interventions: Behavioral: Compass for Care (Well-being intervention)
- Compass for Care (Safety intervention) (Active Comparator): Participants receive 12 weekly modules and tailored messages delivered via text message or email. The intervention focuses on safety behaviors (e.g., weather safety, first aid, home safety, etc.)
  Interventions: Behavioral: Compass for Care (Safety intervention)

INTERVENTIONS:
Behavioral: Compass for Care (Well-being intervention) — Participants receive 12 weekly modules containing interactive activities and static content and tailored messages delivered via text message or email. The intervention focuses on five self-care behaviors critical to ADRD caregiver well-being: 1) taking time to recharge; 2) finding information about your loved one's diagnosis and needs; 3) discovering your strengths and limits; 4) exploring outside help; and 5) seeking emotional support.
  Arms: Compass for Care (Well-being intervention)
Behavioral: Compass for Care (Safety intervention) — Participants receive 12 weekly modules and tailored messages delivered via text message or email. The intervention focuses on safety behaviors (e.g., weather safety, first aid, home safety, etc.)
  Arms: Compass for Care (Safety intervention)

SUMMARY:
In the US, the over 11 million Americans currently providing unpaid care to a family member, relative, or friend with Alzheimer's disease or a related dementia (ADRD) are over 6 times more likely than the general population to suffer from depression (33.9% vs. 5%), and nearly 60% rate their emotional distress as high or very high. The purpose of this Phase II research is to continue the successful work of the pilot development and testing by conducting a rigorous scientific study of the effects of Compass for Care, a digital program that customizes behavior change guidance for using five self-care behaviors critical to ADRD caregiver well-being: 1) taking time to recharge; 2) finding information about your loved one's diagnosis and needs; 3) discovering your strengths and limits; 4) exploring outside help; and 5) seeking emotional support.

DETAILED DESCRIPTION:
The efficacy of the Compass for Care intervention is being tested in a randomized trial involving up to 305 caregivers caring for a family member or friend with Alzheimer's disease or a related dementia (ADRD). Caregivers who meet study inclusion criteria (e.g., being an ADRD caregiver caring for a family member or friend for 8+ hours/week, residing in the US, agreeing to receive daily text or email messages for three months, not indicating suicidal ideation, and experiencing a level of caregiver burden) as assessed in on online screening survey, are invited to participate in the study.

Caregivers are randomly assigned to either the treatment or attention control condition. The treatment group is provided access to the 12-week Compass for Care mobile first program and attention control group is provided access to a 12-week mobile optimized intervention focused on safety behaviors. Both interventions are delivered in weekly modules and include daily messages delivered by email or text message.

Follow-up assessments are conducted online at 3, 6, and 9 months. Outcomes include caregiver burden, depression, perceived stress, emotional and physical health, life satisfaction, resilience, and well-being. Study protocols include best practices for maximizing retention at follow-up in research.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and speak English
2. Aged 18+
3. Residing in the U.S.
4. Regularly use the internet
5. Agree to receive daily messages by email or text during the 3-month intervention period
6. Currently providing at least 8 hours of unpaid care to a family member or friend diagnosed with Alzheimer's disease, Lewy body dementia, frontotemporal dementia, vascular dementia, dementia type not specified, or mixed dementia
7. Have been providing care for at least 3 months;
8. Score of 3 or higher on the Zarit burden item (Overall, how burdened do you feel in caring for your relative) OR a score of 2 on this item and a score of 2+ on the PHQ-2 assessment (i.e., Little interest or pleasure in doing things; Feeling down, depressed, or hopeless)
9. Expecting to provide care to their family member or friend for at least three more months, or don't know how much longer they will be providing care

Exclusion Criteria:

1. Indicating suicidal ideation based upon the PHQ-9 suicidality ideation item (i.e., Thoughts that you would be better off dead, or of hurting yourself)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Zarit Burden Interview (ZBI) | Baseline, 3, 6, and 9 months' follow-up
  Developed from the 29 and 22-item versions, this shortened 12-item Zarit Burden Interview measure assesses subjective burden among caregivers of individuals with dementia. Caregivers are asked to rate items (e.g., Do you feel… that your health has suffered because of your involvement with your relative?) on a 5-point scale with 0 = never to 4 = nearly always. Cronbach's alpha is .88.

SECONDARY OUTCOMES:
Patient Health Questionaire (PHQ-9) | Baseline, 3, 6, and 9 months' follow-up
  Depression is being assessed using the PHQ-9, which asks the number of days in the past two weeks the respondent had experienced each of the Diagnostic and Statistical Manual (DSM) symptoms of depression, minus suicidality. Response options are 0 = Not at all, 1 = Several days, 2 = More than half the days, and 3 = Nearly every day. Scores are summed to produce a total score, and a PHQ-9 cutpoint ≥ 10 is used to define moderate to severe depression. Both depression symptoms (i.e., total score) and prevalence of current depression (score > 10) will be examined in this study.
Resilience Evaluation Measure (REM-3) | Baseline, 3, 6, and 9 months' follow-up
  Developed by ProChange, this 3-item survey assesses three key drivers of resilience: mindset, meaning, and social connections. Items are rated on a 5-point scale with 1 = never, 2 = rarely, 3 = sometimes, 4 = often, and 5 = almost always. Cronbach's alpha is .81.
World Health Organization Well-Being Index (WHO-5) | Baseline, 3, 6, and 9 months' follow-up
  The WHO-5 is a widely used measure that assesses well-being. Respondents are asked to rate five items (e.g., I have felt calm and relaxed) in relation to how they've felt over the last two weeks. Responses range on a 6-point scale from 0=At no time to 5=All of the time.
Cohen's Perceived Stress | Baseline, 3, 6, and 9 months' follow-up
  Originally developed in 1983, the Perceived Stress Scale (PSS) includes 10 items (e.g., In the last month, how often have you felt that you were unable to control the important things in your life) focused on varied situations. Respondents rate the items on a 5-point scale ranging from 0 = never to 4 = very often.
Perceived Change Index | Baseline, 3, 6, and 9 months' follow-up
  This measure of well-being assesses factors associated with increased risk for adverse emotional and physical outcomes among caregivers. Caregivers are asked to rate 13 items (e.g., ability to manage day to day) on a 5- point scale with 1 = became much worse to 5 = improved a lot over the past month. Negatively worded items are reversed scored and an overall measure mean is computed. Cronbach's alpha is .88.
Cantril/Gallup Life Evaluation Index | Baseline, 3, 6, and 9 months' follow-up
  In its World Poll administered in 150 countries, Gallup, Inc. uses the 2-item Cantril Self-Anchoring Scale and a simple scoring algorithm to assess subjective well-being. Respondents are asked to rate their current life-and then to rate their future life, "say about five years from now"-on a ladder where 0 represents the worst possible life and 10 best possible life. Individuals who rate their current life a "7" or higher AND their future life an "8" or higher are classified as "thriving." Individuals who rate their current and future lives a "4" or lower are classified as "suffering." All others are "struggling." Previous research has shown that those classified as thriving experience less depressive symptoms, higher physical and emotional health and have fewer health risk behaviors than those in struggling and suffering.

CONTACTS AND LOCATIONS:
Overall Officials: Kerry E Evers, PhD, Study Director — Pro-Change Behavior Systems
Locations (1):
- Pro-Change Behavior Systems, Narragansett, Rhode Island, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT06249139/ICF_000.pdf